CLINICAL TRIAL: NCT02864706
Title: 5, 6 or 7 Year Follow-up Control After the SCHEDULE Study (SCANDINAVIAN HEART TRANSPLANT EVEROLIMUS DE NOVO STUDY WITH EARLY CNI AVOIDANCE)
Brief Title: SCHEDULE Follow Up Visit 5-7 yr
Acronym: CRAD001ANO05
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ANO05; CRAD001ANO026YFU (Other: Novartis Pharmaceuticals); 2016-000404-28 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-08-12 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Heart Transplantation
Keywords: allograft rejection; xenograft rejection; host vs graft disease; transplant
MeSH Terms: conditions — Graft vs Host Disease | interventions — Everolimus; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVEROLIMUS (Experimental): patients received everolimus (Certican), low-exposure CsA (Neoral), mycophenolate mofetil (MMF) and corticosteroids with CsA withdrawal after 7-11 weeks
  Interventions: Drug: Everolimus
- Control (Active Comparator): patients received standard CsA, MMF and corticosteroids
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Corticosteroids

INTERVENTIONS:
Drug: Everolimus — All patients, independent of their initial randomization in the core study, were followed up as in one single group
  Commercially available everolimus (Certican®), oral route, was used.
  Arms: EVEROLIMUS
Drug: Cyclosporine — Cyclosporine (CsA) control group target blood level: 150-350 ng/mL (month 1-3); 100-250 ng/mL (month 4-6); 60-200 ng/mL (month 7-12); everolimus group target blood level: 75-175 ng/mL (month 1-3)
  Arms: Control
Drug: Mycophenolate mofetil — Mycophenolate mofetil (MMF) target dose for control group: 2000-3000 mg/day everolimus group target dose: 1500-2000 mg/day and 75-175 ng/mL after week 11
  Arms: Control
Drug: Corticosteroids — Corticosteroids (CS) initiated at 0.2-0.5 mg/kg/day. Tapered to no less than 0.1 mg/kg at Month 3 for control and everolimus groups.
  Arms: Control

SUMMARY:
The major aim of this extension study was to evaluate the long-term effect (i.e. 5 to 7 years) of early initiation of everolimus and early elimination of CsA compared to standard immunosuppressive regimen including CsA on primary and secondary endpoints investigated in the SCHEDULE (NCT01266148) main study.

DETAILED DESCRIPTION:
This protocol was written to describe the procedures for a single 5, 6 or 7 year follow-up control visit of patients who participated in the 12-month SCHEDULE (NCT01266148) study and the following 3-year follow-up examination/visit. The aim of this 5 to 7-year follow-up visit was to examine the effect of long term treatment, i.e. 5, 6 or 7 years, with early initiation of everolimus (Certican®) and early elimination of cyclosporine (CsA), compared to standard immunosuppressive regimen including CsA, on renal and heart function. During the time period of this follow-up examinations, this visit was performed as part of a routine annual visit 5, 6 or 7 years since transplantation (and inclusion in the original SCHEDULE study).

Study code of SCHEDULE, the core study: CRAD001ANO02 (EudraCT No.: 2009-013074-41)

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in the SCHEDULE 12-month main study, and who completed the 3 year follow-up visit
* Patients who are coming for a regular annual clinic visit 5 to 7 years after randomization in the main study
* Obtaining of a separate signed patient informed consent will be required for participation in this follow-up examination.

Exclusion Criteria:

* Patients with a retransplanted heart since the original SCHEDULE study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Denmark (2):
  - Novartis Investigative Site, Århus N
  - Novartis Investigative Site, Copenhagen
- Novartis Investigative Site, Oslo, Norway
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Andreassen AK, Andersson B, Gustafsson F, Eiskjaer H, Radegran G, Gude E, Jansson K, Solbu D, Karason K, Arora S, Dellgren G, Gullestad L; SCHEDULE investigators. Everolimus Initiation With Early Calcineurin Inhibitor Withdrawal in De Novo Heart Transplant Recipients: Three-Year Results From the Randomized SCHEDULE Study. Am J Transplant. 2016 Apr;16(4):1238-47. doi: 10.1111/ajt.13588. Epub 2016 Jan 28. PMID 26820618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 95 patients (48 everolimus, 47 controls), attended the follow-up visit at 5-7 years post-transplant and were included in the safety population
  The PP population (27 everolimus, 35 controls) excluded 7 patients in the everolimus group and 11 in the control group who discontinued study drug prematurely
Pre-assignment Details: Two patients randomized to everolimus did not provide a month 12 measured GFR (mGFR) value and were excluded from the ITT population, which thus comprised 93 patients (46 everolimus, 47 controls).
Period: Overall Study
Arm/Group | Everolimus | Control
Started | 48 | 47
Safety Set | 48 | 47
Intent to Treat | 46 | 47
Completed | 48 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat Set (ITT Set) consists of patients who:
  * were included in the ITT in the Clinical Study Reports Addendum dated 11 August 2015 for the 3 year Follow-up visit
  * had at least one assessment of the efficacy variables mGFR or cGFR at the 5 to 7 year Follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Control | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.13 (13.43) | 52.11 (11.61) | 51.11 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Set
  Participants
    Female | 13 | 12 | 25
    Male | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 47 | 44 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Measured Glomerular Filtration Rate (mGFR)
Description: Renal function as assessed by measured Glomerular Filtration Rate (mGFR) (Cr-EDTA or iohexol clearance). Baseline Visit 1 and Patient 4252 excluded from the intent treat analysis set.
Time Frame: at the 5-7 year follow-up visit
Population: intent to treat. 1 patient was excluded from ITT due to missing mGFR.
Measure: Least Squares Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 45 | 46
mL/min/1.73m2 | 74.7 (23.3) | 62.4 (16.5)
Statistical Analysis 1: Comparison: Everolimus vs Control; Test type: Superiority; p = 0.0043, ANCOVA; Incidence of CAV at 5-7 yrs was compared between groups using Cochran-Mantel-Haenszel test with stratification according to baseline distribution

2. Secondary Outcome: Progression of Cardiac Allograft Vasculopathy (CAV) Recorded by Intravascular Ultrasound (IVUS)
Description: Cardiac Allograft Vasculopathy (CAV) was defined as mean maximal intimal thickness (MIT)
  ≥0.5 mm, measured for the entire matched pullback recording by intravascular ultrasound (IVUS). The incidence of CAV at 5-7 years was compared between groups using the Cochran-Mantel-Haenszel test with stratification according to baseline distribution of CAV incidence.
Time Frame: within 5-7 years
Population: Intent to Treat.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 36 | 35
mm | 0.13 (0.15) | 0.23 (0.24)
Statistical Analysis 1: Comparison: Everolimus vs Control; Test type: Superiority; p = 0.037, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percent of Participants With Incidence of Coronary Allograft Vasculopathy (CAV)
Description: as for outcome 2
Time Frame: at the 5-7 year follow-up
Population: Intent to Treat
Measure: Number; unit: percent of participants
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 36 | 35
percent of participants | 53 | 74

4. Secondary Outcome: Myocardial Structure and Function
Description: Myocardial structure and function by echocardiography assessment measured by ventricular end systolic diameter.
Time Frame: within 5-7 years
Population: intent to treat
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 47
cm
  LVESD (left ventricular end systolic diameter): number analyzed (Participants) | 35 | 39
  LVESD (left ventricular end systolic diameter) | 3.1 (0.8) | 3.1 (0.6)
  LVEDD (left ventricular end diastolic diameter): number analyzed (Participants) | 44 | 46
  LVEDD (left ventricular end diastolic diameter) | 4.7 (0.6) | 4.9 (0.6)

5. Secondary Outcome: Quality of Life by SF-36 Change From Pre-transplantation to 5-7 Year Follow-up
Description: This Quality of life Short Form Survey with 36 items (Minnesota Living with Heart Failure Questionnaire)was administered to patients pre-transplantation and after transplantation at the 5-7 year visit. This data represents the change. The survey consist of scores on a scale. Each form is scaled from 0 t 100. 0 = maximum disability and 100 equals no disability.
Time Frame: at the 5-7 year visit
Population: intent to treat
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 47
scores on a scale
  Physical Health Summary: number analyzed (Participants) | 30 | 34
  Physical Health Summary | 16.8 (15.0) | 13.2 (13.3)
  Mental Health Summary: number analyzed (Participants) | 30 | 34
  Mental Health Summary | 10.4 (10.5) | 15.3 (15.5)
  Physical Functioning: number analyzed (Participants) | 35 | 37
  Physical Functioning | 36.7 (38.4) | 40.8 (30.4)
  Role Physical: number analyzed (Participants) | 35 | 37
  Role Physical | 50.2 (32.3) | 55.1 (32.4)
  Bodily Pain: number analyzed (Participants) | 35 | 36
  Bodily Pain | 10.3 (34.8) | 7.2 (34.1)
  General Health: number analyzed (Participants) | 37 | 38
  General Health | 25.7 (26.4) | 23.4 (25.6)
  Vitality: number analyzed (Participants) | 33 | 37
  Vitality | 30.0 (25.8) | 28.9 (29.0)
  Social Functioning: number analyzed (Participants) | 36 | 37
  Social Functioning | 39.9 (31.5) | 43.9 (32.4)
  Role Emotional: number analyzed (Participants) | 36 | 37
  Role Emotional | 23.8 (36.7) | 42.8 (46.5)
  Mental Health: number analyzed (Participants) | 33 | 37
  Mental Health | 8.6 (17.2) | 14.4 (25.8)

6. Secondary Outcome: Change From Baseline in the Euro Quality of Life 5D
Description: Change from baseline in Euro Quality of Life-5D from 3 Year Follow-Up to 5 to 7 Year Follow-Up Baseline Visit 1 (ITT Set)
  Euro Quality of Life 5D (EQ-5D): is a descriptive system of healthrelated quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) each of which can be assessed as one of three levels of severity (no problems/some or moderate problems/extreme problems). A Visual Analogue Scale (VAS)-scale is also included in the EQ-5D questionnaire.
  The EQ-5D index is calculated based on the United Kingdom Time Trade-Off (TTO) N3 value set which converts the five dimensions scores into a single measure with a possible range from -0.163 (worst possible health state) to +1 (perfect health). A positive change from baseline indicates an improvement in Quality of Life.
Time Frame: Baseline, 5-7 year visit
Population: intent to treat
Measure: Mean (Standard Deviation); unit: scores on the scale
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 46
scores on the scale | 0.2323 (0.3849) | 0.2982 (0.3274)

7. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS)
Description: Change in visual analog scale (VAS) from baseline to the 5 to 7 Year follow up visit.
  0 is no pain; and 10 is the worst possible pain
Time Frame: baseline, at the 5-7 year visit
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 47
mm | 35.6 (26.9) | 34.0 (32.0)

8. Secondary Outcome: Number of Participants With Beck Depression Inventory (BDI)
Description: Beck Depression Inventory (BDI) Score has the following categories of depression. Normal, Mild, Moderate Severe and Missing.
Time Frame: at the 5-7 year visit
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 47
Participants
  Normal | 15 | 13
  Mild | 6 | 4
  Moderate | 2 | 5
  Severe | 1 | 0
  Missing | 3 | 5

ADVERSE EVENTS:
Time Frame: An average of 3 years (from the 3 year follow-up visit to the 5-7 year follow-up visit)
Groups:
- Everolimus: All participants who were included in the initial core study SCHEDULE (CRAD001ANO02) who received an immunosuppressive regimen consisting of CsA, MMF and CS throughout the study.
Arm/Group | Everolimus | Control
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 26/48 | 18/47
Other Adverse Events (participants affected / at risk) | 15/48 | 4/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=48) | Control (N=47)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Heart transplant rejection (Immune system disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 3
Sepsis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus (N=48) | Control (N=47)
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Oedema peripheral (General disorders) | 5 | 0
Pneumonia (Infections and infestations) | 8 | 2
Sepsis (Infections and infestations) | 3 | 0

LIMITATIONS AND CAVEATS:
There is no investigational medicinal product (IMP). This study is a single follow-up visit. Hence patients' first and last visit dates are the same.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02864706/SAP_000.pdf
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT02864706/Prot_001.pdf